CLINICAL TRIAL: NCT06454968
Title: Orelabrutinib Combined With Obinutuzumab and Lenalidomide (OGL Regimen) as First-line Treatment for Marginal Zone Lymphoma：a Multicenter Prospective Single Arm Trial
Brief Title: Orelabrutinib Combined With Obinutuzumab and Lenalidomide (OGL Regimen) as First-line Treatment for Marginal Zone Lymphoma.
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Peking Union Medical College Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: PUMCH-NHL-017
Record Dates: First submitted 2024-05-27; First posted 2024-06-12 (Actual); Last update posted 2024-06-18 (Actual); Status verified 2024-05

CONDITIONS: Marginal Zone Lymphoma
Keywords: Orelabrutinib; Marginal Zone Lymphoma; obinutuzumab; lenalidomide
MeSH Terms: conditions — Lymphoma, B-Cell, Marginal Zone | interventions — orelabrutinib; obinutuzumab; Lenalidomide

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- OGL (Experimental): Orelabrutinib: 150mg qd d1-d21/C1-C6 obinutuzumab: 1000mg iv d1,d8,d15/c1, 1000mg iv d1/C2-C6 lenalidomide：25mg po qd d1-14/C1-C6 Orelabrutinib: 150mg qd d1-d28/C7-C12
  Interventions: Drug: Orelabrutinib, obinutuzumab, lenalidomide

INTERVENTIONS:
Drug: Orelabrutinib, obinutuzumab, lenalidomide — Orelabrutinib: 150mg qd d1-d21/C1-C6 obinutuzumab: 1000mg iv d1,d8,d15/c1, 1000mg iv d1/C2-C6 lenalidomide：25mg po qd d1-14/C1-C6 Orelabrutinib: 150mg qd d1-d28/C7-C12

SUMMARY:
This is a multicenter prospective single arm phase II study, and the purpose of this study is to evaluate the safety and efficacy of orelabrutinib combined with obinutuzumab and lenalidomide in untreated marginal zone lymphoma. The primary objective was the best complete response rate (CRR).

DETAILED DESCRIPTION:
Marginal zone lymphomas (MZL) are a type of lymphoma that originates from the marginal zone tissue of the lymphoid follicles (Mucosa-associated lymphoid tissue, MALT), and include three subtypes: MALT lymphoma, nodal MZL, and splenic MZL. The incidence of MZL is second only to diffuse large B-cell lymphoma (DLBCL) and follicular lymphoma (FL), accounting for approximately 7.8% of all non-Hodgkin lymphomas (NHL). MZL is considered an indolent lymphoma, with patients generally having a better overall survival prognosis. Despite this, some patients still face the challenges of disease relapse or transformation into large cell lymphoma, leading to a poor prognosis.

We conduct this prospective, phase II, single-arm clinical study to initially explore the efficacy and safety of Orelabrutinib combined with obinutuzumab and lenalidomide in patients with previously untreated marginal zone lymphoma. The patients will be treated with 6 cycles of OGL regimen. Patients with CR/PR after 6 cycles of OGL treatment will be treated with 6 cycles of single-agent orelabrutinib regimen.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years, either sex.
* Histopathologically confirmed B-cell non-Hodgkin lymphoma MZL (splenic, nodal, or extra-nodal).
* At least 1 measurable lesion
* Eligible for treatment: meets the GELF criteria, or has clinical symptoms/organ dysfunction related to the disease
* Patients who are not suitable for local radiotherapy or whose condition progresses after local treatment, and those not suitable for local radiotherapy include the following situations:

  * Ann Arbor non-continuous Stage II or Stage III-IV non-gastric MALT and nodal MZL
  * SMZL (Splenic Marginal Zone Lymphoma)
  * Gastric MALT with Lugano Stage II2/IIE/IV
* ECOG performance status (PS) score of 0-2.
* Expected survival time is ≥3 months
* Sign the Informed consent

Exclusion Criteria:

* Currently has other malignant tumors;
* Lymphoma involving the central nervous system
* Allergic to any of the study drugs;
* Active infection or uncontrolled HBV infection (DNA>105/ml), HIV/AIDS, or other severe infectious diseases;
* Pregnant or lactating women and women of childbearing age who are unwilling to use contraception;
* Any other conditions deemed unsuitable for participation in this trial by the investigator.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 45 (Estimated)
Dates: Start 2024-06-20 (Estimated); Primary Completion 2026-06-01 (Estimated); Study Completion 2028-06-01 (Estimated)

PRIMARY OUTCOMES:
the best complete response rate | At the end of cycle 12(the first 6 cycles are 21 days each, and the following 6 cycles are 28 days each)
  CRR is defined as the proportion of patients with a best response of CR

SECONDARY OUTCOMES:
ORR | At the end of therapy(up to 42 weeks)
  ORR is defined as the proportion of patients with a response of CR or PR
CRR | At the end of therapy(up to 42 weeks)
  CRR is defined as the proportion of patients with a best response of CR
The best ORR | At the end of cycle 12(the first 6 cycles are 21 days each, and the following 6 cycles are 28 days each)
  The best ORR is defined as the proportion of patients with a best response of CR or PR
2 years progression-free survival Progression free survival (PFS) | From date of signing the informed consent until the date of first documented progression or date of death from any cause, whichever came first, assessed up to 2 years]
  PFS is defined as the time from registration to the first occurrence of progression or relapse as assessed by the investigator, or death from any cause. PFS for patients without disease progression, relapse, or death will be censored at the time of the last tumor assessment.
2 years overall survival | From date of signing the informed consent until the date of death from any cause, whichever came first, assessed up to 2 years]
  Overall survival is defined as the period from the induction registration to death from any cause. Patients who have not died until the time of the analysis will be censored at their last contact date.
TTR | Up to 2 years
  TTR is defined as the time from registration to the first response.
Duration of Response (DOR) | Up to 2 years
  Duration of response as defined as the period from the first response (at least PR) to treatment until evidence of disease progression, relapse or death of any cause. Patients alive without progression and relapse will be censored at the latest tumor assessment date or the stopping date.
The occurrence of adverse events and serious adverse events | One month after the end of treatment（up to 46 weeks）
  Adverse events will be graded by the investigator according to the NCI-CTCAE Version 5.0.

CONTACTS AND LOCATIONS:
Locations (1):
- Peking Union Medical College Hospital, Beijing, Beijing Municipality, China